CLINICAL TRIAL: NCT01041807
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy Profile of COZAAR XQ in Usual Practice
Brief Title: Cozaar XQ Re-examination Study (MK-0954-349)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0954-349; 2009_004 (Other: Merck Registration Number)
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — amlodipine-losartan drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Participants with hypertension treated with amlodipine/losartan(Cozaar XQ)
  Interventions: Drug: amlodipine/losartan

INTERVENTIONS:
Drug: amlodipine/losartan — amlodipine/losartan (COZAAR XQ) prescribed according to the current local label
  Other Names: COZAAR XQ

SUMMARY:
This survey is conducted for preparing application material for re-examination under the Pharmaceutical Affairs Law and its Enforcement Regulation; its aim is to reconfirm the clinical usefulness of COZAAR XQ through collecting the safety and efficacy information according to the Re-examination Regulation for New Drugs.

ELIGIBILITY:
Inclusion criteria:

* Participant with essential hypertension
* Participant who is treated with COZAAR XQ within local label for the first time

Exclusion criteria:

* Participant who is treated with COZAAR XQ before contract and out of enrollment period
* Participant who has a contraindication to COZAAR XQ according to the local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with essential hypertension not adequately controlled with amlodipine or losartan monotherapy; initial therapy for participants with stage 2 hypertension
Sampling Method: Probability Sample
Enrollment: 669 (Actual)
Dates: Start 2010-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with any adverse experience | Up to 14 days after last treatment
Change of sitting systolic and diastolic blood pressure (SiSBP, SiDBP) after treatment and overall efficacy evaluation by investigator | At 8 weeks after first treatment

SECONDARY OUTCOMES:
Change of sitting systolic and diastolic blood pressure (SiSBP, SiDBP) after treatment and overall efficacy evaluation by investigator | At 24 weeks after first treatment